CLINICAL TRIAL: NCT00024362
Title: A Phase II Trial of BBR 3464 as First Line Treatment in Patients With Inoperable, Locally Advanced or Metastatic Adenocarcinoma of the Pancreas
Brief Title: BBR 3464 in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer That Cannot be Treated With Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068924; THERADEX-TPT-II-06; NOVUSPHARMA-TPT-II-06
Record Dates: First submitted 2001-09-13; First posted 2004-02-06 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — BBR 3464

INTERVENTIONS:
Drug: BBR 3464

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BBR 3464 in treating patients who have locally advanced or metastatic pancreatic cancer that cannot be treated with surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall survival of patients with inoperable locally advanced or metastatic adenocarcinoma of the pancreas treated with BBR 3464. II. Determine the response rate, duration of response, time to disease progression, and duration of stable disease in patients treated with this drug. III. Determine the incidence and severity of the toxic effects of this drug in these patients. IV. Determine the disease-related symptoms in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive BBR 3464 IV over 1 hour on day 1. Treatment repeats every 21 days for a minimum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 9 weeks.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed adenocarcinoma of the pancreas Inoperable locally advanced or metastatic disease Previously untreated disease At least 1 measurable lesion Lesions in a previously irradiated field are not considered measurable Brain metastases allowed provided symptoms are stable and patient is receiving a stable dose of steroids within 1 month prior to study

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN ALT or AST no greater than 2 times ULN (5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No congestive heart failure No angina pectoris (even if medically controlled) No myocardial infarction within the past year No uncontrolled hypertension No arrhythmia Neurologic: No significant neurological disorder except that caused by metastatic disease or psychiatric disorders No clinically significant abnormal findings on audiogram or neurological examination Other: No other serious illness or medical condition No uncontrolled concurrent infection No prior disposition to diarrhea (e.g., Crohn's disease or ulcerative colitis) No poor nutritional status that would be compromised by severe diarrhea No other prior or concurrent malignancy except: Curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix OR Other cancer curatively treated by surgery alone that has not recurred for more than 5 years No other condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy No concurrent antitumor immunotherapy Chemotherapy: No prior chemotherapy No other concurrent antitumor chemotherapy Endocrine therapy: See Disease Characteristics No prior endocrine therapy No concurrent antitumor hormonal therapy Radiotherapy: See Disease Characteristics Prior single fraction of radiotherapy for palliation allowed No concurrent radiotherapy except for local palliation to a nontarget lesion Surgery: See Disease Characteristics Prior surgeries allowed At least 4 weeks since prior major thoracic and/or abdominal surgery (2 weeks for biliary drainage procedures) and recovered Other: At least 30 days since prior investigational drugs No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05

CONTACTS AND LOCATIONS:
Overall Officials: George L. Miller, MD, Study Chair — Oklahoma Oncology, Incorporated at LaFortune Cancer Center
Locations (9):
- United States (9):
  - Arizona Oncology Associates, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oklahoma Oncology Inc., Tulsa, Oklahoma
  - Boston Baskin Cancer Group, University Tennessee Oncology/Hematology Group, Memphis, Tennessee
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Massey Cancer Center, Richmond, Virginia